CLINICAL TRIAL: NCT05936502
Title: Ascertaining the Radiologic Prognostic Importance of Extranodal Extension on Imaging (iENE) in Head and Neck Cancer Part of the Evaluation Prognostic and Predictive Indicators in Head and Neck Cancer (EPIC) Programme, Run Under the Auspices of the Head and Neck Inter Group (HNCIG, Www.Hncig.Org)
Brief Title: Ascertaining the Radiologic Prognostic Importance of Extranodal Extension on Imaging (iENE) in Head and Neck Cancer
Acronym: EPIC-iENE DATA
Status: Completed | Type: Observational
Sponsor: Head and Neck Cancer International Group (Other)
Responsible Party: Principal Investigator, Professor Hisham Mehanna, Professor, Head and Neck Cancer International Group
Other Study IDs: EPIC-iENE DATA
Record Dates: First submitted 2023-05-24; First posted 2023-07-07 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Extranodal Extension; Human Papilloma Virus Related Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Extranodal Extension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Extranodal extension — Extranodal extension presence or absence on radiology and pathology assessment

SUMMARY:
Extranodal extension (ENE) refers to the spread of head and neck squamous cell carcinoma (HNSCC) outside the lymph nodes. It is a well-known factor that indicates a poorer prognosis and outcome for patients who have undergone surgical removal of the cancer. In such cases, it is recommended to combine chemotherapy with radiation therapy after surgery.

As the number of cases of HNSCC related to the human papillomavirus (HPV) is increasing, treatment approaches have shifted towards using radiation therapy as the primary treatment method instead of surgery. This raises an important question about the significance of ENE observed through imaging tests (referred to as iENE) and its impact on the prognosis. Unfortunately, this question remains unanswered.

The objective of this project is to conduct a comprehensive study across multiple medical institutions. The investigators will gather data including scan results, histopathology reports, and data from patient charts from individuals who have been treated for head and neck cancer. The aim is to analyze and correlate the findings between the pathological evidence of ENE and the imaging results, while also assessing the prognostic value of iENE. Additionally, the investigators will explore the influence of HPV status on these factors.

By collecting and analyzing this data, the investigators hope to establish standardized criteria that can assist radiologists in accurately identifying ENE through imaging tests. This research is essential for enhancing our understanding of HNSCC and improving the effectiveness of diagnostic procedures and treatment planning.

ELIGIBILITY:
Inclusion Criteria:

The investigators will examine data from consecutive patients at each site treated between 1/1/1999 and 12/31/2020. Patients must fulfil all these criteria:

i. Been treated for oral cavity, oropharyngeal, carcinoma of unknown primary, laryngeal, or hypopharyngeal squamous cell carcinoma and be over the age of 18.

ii. The participants must have been treated with curative intent via surgery, radiotherapy, or chemoradiotherapy or a combination within the study inclusion period.

iii. The participants must have had CT or/and MRI scans of the neck, performed within 12 weeks before the start of treatment.

iv. Results for the presence or absence of extranodal extension on CT or/and MRI scans, or ability to report them within the deadline period.

v. For surgically-treated patients: Results for the presence or absence of both extranodal extension on histopathology and on radiology, or ability to report them within the deadline period.

vi. Must have had at least two years of follow-up, or death. vii. Data on staging must be available at least in TNM 7th edition or later editions.

Exclusion Criteria:

i. Patients who were diagnosed with distant metastasis at presentation. ii. Patients treated palliatively at first presentation iii. Patients presenting with recurrent disease who don't meet all the eligibility criteria above

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented and treated for Head and neck squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
To assess the accuracy of the identification of iENE by radiologists in real world situations by correlating with histopathology (pENE) | 31 December 2023
  Endpoints: Accuracy of a radiologic "call" of iENE (with pENE being the gold standard comparator) by radiologists not trained for any standardized diagnostic classification systems for iENE.
To evaluate the prognostic significance (overall survival rates) of iENE. | 31 December 2023
  Endpoints: Overall survival rates based on presence of iENE and pENE
To evaluate the prognostic significance (recurrence rates) of iENE | 31 December 2023
  Endpoints: Recurrence rates based on presence of iENE and pENE
To evaluate the prognostic significance (overall survival rates) of iENE: Risk stratify HNSCC patients based on presence of radiographic ENE, according to their HPV status and N stage | 31 December 2023
  Endpoints: Overall survival rates based on presence of various degrees of iENE and pENE
To evaluate the prognostic significance (recurrence rates) of iENE: Risk stratify HNSCC patients based on presence of radiographic ENE, according to their HPV status and N stage | 31 December 2023
  Endpoints: Recurrence rates based on presence of various degrees of iENE and pENE

SECONDARY OUTCOMES:
Improve the diagnosis of iENE: Determine radiological features of iENE that best correlate with pENE (the gold standard comparator) | 31 December 2023
  Endpoints: Diagnostic accuracy of various radiographic features of iENE with pENE.
Assess the utility of various existing standardized diagnostic classification systems in accurately diagnosing iENE | 31 December 2023
  Endpoints: Diagnostic accuracy of published standardized classification systems with pENE
Measure interobserver variability amongst radiologists in grading radiographic ENE and to measure impact of standardized criteria on this variability | 31 December 2023
  Endpoints: Interobserver variability measured by Cohen's kappa

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Mehanna, PhD, Principal Investigator — University of Birmingham; Christina Henson, MD, Principal Investigator — The University of Oklahoma Health Sciences Center; Ahmad K. Abou-Foul, MD, Principal Investigator — University of Birmingham; Paul C Nankivell, PhD, Principal Investigator — University of Birmingham
Locations (12):
- United States (3):
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Mount Sinai Health System, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Royal Adelaide Hospital, Adelaide, Australia
- Copenhagen University Hospitals, Copenhagen, Denmark
- Georges Pompidou European Hospital, Paris, France
- Germany (2):
  - University of Cologne, Cologne
  - Technical University of Munich, Munich
- Catalan Institute of Oncology, Barcelona, Spain
- University Hospital Zürich, Zurich, Switzerland
- United Kingdom (2):
  - University Hospitals Birmingham, Birmingham
  - Leeds Teaching Hospitals NHS Trust, Leeds

IPD SHARING:
Plan to Share IPD: Undecided
The data will bill kept in the HNCIG database, and might be shared with other researchers following a reasonable request (and following agreement by the HNCIG board)